CLINICAL TRIAL: NCT03564340
Title: A Phase 1/2 Study of REGN4018 (Ubamatamab), a MUC16×CD3 Bispecific Antibody, Administered Alone or in Combination With Cemiplimab in Patients With Recurrent Ovarian Cancer or Other Recurrent MUC16+ Cancers
Brief Title: Study of REGN4018 (Ubamatamab) Administered Alone or in Combination With Cemiplimab in Adult Patients With Recurrent Ovarian Cancer or Other Recurrent Mucin-16 Expressing (MUC16+) Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R4018-ONC-1721; 2024-510783-23-00 (EU CTIS Number); 2019-003298-24 (EudraCT Number)
Record Dates: First submitted 2018-05-17; First posted 2018-06-20 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Ovarian Cancer; Recurrent Fallopian Tube Cancer; Recurrent Primary Peritoneal Cancer; Recurrent Endometrial Cancer; Endometrial Cancer; Low-grade Serous Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Endometrial Neoplasms | interventions — cemiplimab; sarilumab; tocilizumab; Biosimilar Pharmaceuticals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy (Experimental): REGN4018 administration
  Interventions: Drug: Ubamatamab; Drug: Sarilumab; Drug: Tocilizumab
- Combination Therapy (Experimental): REGN4018 and cemiplimab administration
  Interventions: Drug: Ubamatamab; Drug: Cemiplimab

INTERVENTIONS:
Drug: Ubamatamab — Administered per the protocol
  Other Names: REGN4018
Drug: Cemiplimab — Administered per the protocol
  Other Names: REGN2810; Libtayo®
  Arms: Combination Therapy
Drug: Sarilumab — Administered per the protocol
  Other Names: Kevzara®; REGN88; SAR153191
  Arms: Monotherapy
Drug: Tocilizumab — Administered per the protocol
  Other Names: ACTEMRA®; Biosimilar
  Arms: Monotherapy

SUMMARY:
The main purpose of this study is to:

* Learn about the safety of ubamatamab and to find out what dose of ubamatamab can be given alone or with cemiplimab to patients with ovarian cancer or cancer of the uterus
* The study will also look at the levels of ubamatamab and/or cemiplimab in the body and measure how well the body can remove the study drug(s). This is called pharmacokinetics
* The study will also look at any signs that ubamatamab alone or with cemiplimab can treat recurrent advanced ovarian cancer or cancer of the uterus
* To find out how safe and tolerable pretreatment is in combination with ubamatamab and to see how well it works to prevent or minimize Cytokine Release Syndrome (CRS)

ELIGIBILITY:
Key Inclusion Criteria:

1. Ovarian Cancer Cohorts Only: Patients with histologically or cytologically confirmed diagnosis of advanced, epithelial ovarian cancer (except carcinosarcoma), primary peritoneal, or fallopian tube cancer who have all of the following:

   1. serum CA-125 level ≥2 x upper limit of normal (ULN) (in screening, not required for low-grade serous carcinoma)
   2. has received at least 1 line of platinum-containing therapy or must be platinum-intolerant (applicable for dose escalation and non-randomized dose expansion cohorts)
   3. documented relapse or progression on or after the most recent line of therapy
   4. no standard therapy options likely to convey clinical benefit
2. Adequate organ and bone marrow function as defined in the protocol
3. Life expectancy of at least 3 months
4. Randomized phase 2 expansion cohort (Ovarian Cancer only): Platinum-resistant ovarian cancer patients who have had 2 to 4 lines of platinum-based therapy as defined in the protocol.
5. Endometrial Cancer Cohorts Only: histologically confirmed endometrial cancer that has progressed or recurrent after prior anti-Programmed Cell Death Ligand 1 (PD-1) therapy and platinum-based chemotherapy:

   1. MUC16 positivity of tumor cells ≥25% by immunohistochemistry (IHC), as defined in the protocol
   2. 1-4 prior lines of systemic therapy, as described in the protocol

Key Exclusion Criteria:

1. Prior treatment with anti-Programmed Cell Death (PD-1)/PD-L1 therapy, as described in the protocol
2. Ovarian Cancer Expansion cohorts only: More than 4 prior lines of cytotoxic chemotherapy (does not apply to low-grade serous ovarian cancer cohort)
3. Prior treatment with a MUC16 - targeted therapy
4. Untreated or active primary brain tumor, central nervous system (CNS) metastases, or spinal cord compression, as described in the protocol
5. History and/or current cardiovascular disease, as defined in the protocol
6. Severe and/or uncontrolled hypertension at screening. Patients taking anti-hypertensive medication must be on a stable anti-hypertensive regimen

Note: Other protocol-defined Inclusion/Exclusion Criteria apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 890 (Estimated)
Dates: Start 2018-05-21 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose-limiting toxicity (DLTs) for ubamatamab monotherapy | From Cycle 1, Day 1 up to 35 days
  Dose Escalation Phase
Number of participants with DLTs for ubamatamab with cemiplimab | From Cycle 2, Day 1 up to 21 days
  Dose Escalation Phase
Number of participants with Treatment-emergent adverse event (TEAE)s (including immune-related adverse events (imAEs)) for ubamatamab monotherapy | Up to 2 years
  Dose Escalation Phase
Number of participants with TEAEs (including imAEs) for ubamatamab with cemiplimab | Up to 2 years
  Dose Escalation Phase
Number of participants with serious adverse events (SAEs) for ubamatamab monotherapy | Up to 2 years
  Dose Escalation Phase
Number of participants with SAEs for ubamatamab with cemiplimab | Up to 2 years
  Dose Escalation Phase
Number of deaths for ubamatamab monotherapy | Up to 2 years
  Dose Escalation Phase
Number of deaths for ubamatamab with cemiplimab | Up to 2 years
  Dose Escalation Phase
Number of participants with laboratory abnormalities (grade 3 or higher per Common Terminology Criteria for Adverse Events [CTCAE]) for ubamatamab monotherapy | Up to 2 years
  Dose Escalation Phase
Number of participants with laboratory abnormalities (grade 3 or higher per CTCAE) for ubamatamab with cemiplimab | Up to 2 years
  Dose Escalation Phase
Concentration of ubamatamab in serum over time for ubamatamab monotherapy | Up to 2 years
  Dose Escalation Phase
Concentration of ubamatamab in serum over time for ubamatamab with cemiplimab | Up to 2 years
  Dose Escalation Phase
Objective response rate (ORR) defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) for ubamatamab monotherapy | Up to 2 years
  Dose Expansion Phase
ORR defined by RECIST 1.1 for ubamatamab with cemiplimab | Up to 2 years
  Dose Expansion Phase

SECONDARY OUTCOMES:
ORR based on RECIST 1.1 for ubamatamab monotherapy | Up to 2 years
  Dose Escalation Phase
ORR based on RECIST 1.1 for ubamatamab with cemiplimab | Up to 2 years
  Dose Escalation Phase
Number of participants with TEAEs (including imAEs) for ubamatamab monotherapy | Up to 2 years
  Dose Expansion Phase
Number of participants with TEAEs (including imAEs) for ubamatamab with cemiplimab | Up to 2 years
  Dose Expansion Phase
Number of participants with SAEs for ubamatamab monotherapy | Up to 2 years
  Dose Expansion Phase
Number of participants with SAEs for ubamatamab with cemiplimab | Up to 2 years
  Dose Expansion Phase
Number of deaths for ubamatamab monotherapy | Up to 2 years
  Dose Expansion Phase
Number of deaths for ubamatamab with cemiplimab | Up to 2 years
  Dose Expansion Phase
Number of participants with laboratory abnormalities (grade 3 or higher per CTCAE) for ubamatamab monotherapy | Up to 2 years
  Dose Expansion Phase
Number of participants with laboratory abnormalities (grade 3 or higher per CTCAE) for ubamatamab with cemiplimab | Up to 2 years
  Dose Expansion Phase
Concentration of ubamatamab in serum over time for ubamatamab monotherapy | Up to 2 years
  Dose Expansion Phase
Concentration of ubamatamab in serum over time for ubamatamab with cemiplimab | Up to 2 years
  Dose Expansion Phase
Change from baseline in quality of life (QoL) as measured by the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 GHS/QoL score for ubamatamab monotherapy | Baseline up to 2 years
  Dose Expansion Phase
  The EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including global health status/quality of life, functional Scales (physical, role, emotional, cognitive, and social) , symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4-point scale, with 1 as "not at all" and 4 as "very much."
Change from baseline in quality of life (QoL) as measured by the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 GHS/QoL score for ubamatamab with cemiplimab | Baseline up to 2 years
  Dose Expansion Phase
Change from baseline in physical functioning as measured by the EORTC QLQ-C30 physical functioning score for ubamatamab monotherapy | Baseline up to 2 years
  Dose Expansion Phase
Change from baseline in physical functioning as measured by the EORTC QLQ-C30 physical functioning score for ubamatamab with cemiplimab | Baseline up to 2 years
  Dose Expansion Phase
Change from baseline in abdominal symptoms as measured by the Measure of Ovarian Symptoms and Treatment (MOST)-Abdominal index score for ubamatamab monotherapy | Baseline up to 2 years
  Dose Expansion Phase excluding the Endometrial Cancer Cohort
  The MOST-24 is a 24-item questionnaire used to measure the impact of chemotherapy on symptoms (21 items) and well-being (3 items). The expected questionnaire completion time is less than 5 minutes.
  The prevalence of each MOST item at assessment time points can be summarized by providing the mean, standard deviation and proportions based on the MOST response format, a numeric rating scale with integers from zero to 10, with five verbal anchors: 'No trouble at all' (0), 'Mild' (1-3), 'Moderate' (4-6), 'Severe' (7-10), and 'Worst I can imagine' (10).
Change from baseline in abdominal symptoms as measured by the MOST-Abdominal index score for ubamatamab with cemiplimab | Baseline up to 2 years
  Dose Expansion Phase Not applicable to Endometrial Cancer Cohort
Time to deterioration in GHS/QoL for ubamatamab monotherapy | Up to 2 years
  Dose Expansion Phase
Time to deterioration in GHS/QoL for ubamatamab with cemiplimab | Up to 2 years
  Dose Expansion Phase
Time to deterioration in physical functioning for ubamatamab monotherapy | Up to 2 years
  Dose Expansion Phase
Time to deterioration in physical functioning for ubamatamab with cemiplimab | Up to 2 years
  Dose Expansion Phase
Time to deterioration in abdominal symptoms for ubamatamab monotherapy | Up to 2 years
  Dose Expansion Phase
Time to deterioration in abdominal symptoms for ubamatamab with cemiplimab | Up to 2 years
  Dose Expansion Phase
Change from baseline in QoL as measured by EQ-5D for ubamatamab monotherapy | Baseline up to 2 years
  Dose Expansion Phase
Change from baseline in QoL as measured by EQ-5D for ubamatamab with cemiplimab | Baseline up to 2 years
  Dose Expansion Phase
ORR based on iRECIST for ubamatamab monotherapy | Up to 2 years
  Dose Escalation and Dose Expansion Phases
ORR based on iRECIST for ubamatamab with cemiplimab | Up to 2 years
  Dose Escalation and Dose Expansion Phases
Best overall response (BOR) based on RECIST 1.1 for ubamatamab monotherapy | Up to 2 years
  Dose Escalation and Dose Expansion Phases
BOR based on iRECIST for ubamatamab monotherapy | Up to 2 years
  Dose Escalation and Dose Expansion Phases
BOR based on RECIST 1.1 for ubamatamab with cemiplimab | Up to 2 years
  Dose Escalation and Dose Expansion Phases
BOR based on iRECIST for ubamatamab with cemiplimab | Up to 2 years
  Dose Escalation and Dose Expansion Phases
Duration of response (DOR) based on RECIST 1.1 for ubamatamab monotherapy | Up to 2 years
  Dose Escalation and Dose Expansion Phases
DOR based on iRECIST for ubamatamab monotherapy | Up to 2 years
  Dose Escalation and Dose Expansion Phases
DOR based on RECIST 1.1 for ubamatamab with cemiplimab | Up to 2 years
  Dose Escalation and Dose Expansion Phases
DOR based on iRECIST for ubamatamab with cemiplimab | Up to 2 years
  Dose Escalation and Dose Expansion Phases
Disease control rate based on RECIST 1.1 for ubamatamab monotherapy | Up to 2 years
  Dose Escalation and Dose Expansion Phases
Disease control rate based on iRECIST for ubamatamab monotherapy | Up to 2 years
  Dose Escalation and Dose Expansion Phases
Disease control rate based on RECIST 1.1 for ubamatamab with cemiplimab | Up to 2 years
  Dose Escalation and Dose Expansion Phases
Disease control rate based on iRECIST for ubamatamab with cemiplimab | Up to 2 years
  Dose Escalation and Dose Expansion Phases
Complete response (CR) rate based on RECIST 1.1 for ubamatamab monotherapy | Up to 2 years
  Dose Escalation and Dose Expansion Phases
CR rate based on iRECIST 1.1 for ubamatamab monotherapy | Up to 2 years
  Dose Escalation and Dose Expansion Phases
CR rate based on RECIST 1.1 for ubamatamab with cemiplimab | Up to 2 years
  Dose Escalation and Dose Expansion Phases
CR rate based on iRECIST 1.1 for ubamatamab with cemiplimab | Up to 2 years
  Dose Escalation and Dose Expansion Phases
Progression-free survival (PFS) based on RECIST 1.1 for ubamatamab monotherapy | Up to 2 years
  Dose Escalation and Dose Expansion Phases
PFS based on iRECIST for ubamatamab monotherapy | Up to 2 years
  Dose Escalation and Dose Expansion Phases
PFS based on RECIST 1.1 for ubamatamab with cemiplimab | Up to 2 years
  Dose Escalation and Dose Expansion Phases
PFS based on iRECIST for ubamatamab with cemiplimab | Up to 2 years
  Dose Escalation and Dose Expansion Phases
Cancer antigen-125 (CA-125) response for ubamatamab monotherapy | Up to 2 years
  Dose Escalation and Dose Expansion Phases
CA-125 response for ubamatamab with cemiplimab | Up to 2 years
  Dose Escalation and Dose Expansion Phases
Presence or absence of anti-drug antibodies against ubamatamab | Up to 2 years
  Dose Escalation and Dose Expansion Phases
Presence or absence of anti-drug antibodies against cemiplimab | Up to 2 years
  Dose Escalation and Dose Expansion Phases

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (51):
- United States (11):
  - University of Alabama_6th Ave, Birmingham, Alabama
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber / Harvard Cancer Center, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University Wexner Medical Center James Comprehensive Cancer Center, Hilliard, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (2):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Peter MacCallum Cancer Center, Melbourne
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Edegem, Antwerp
  - Grand Hopital de Charleroi, Charleroi, Hainaut
  - UZLeuven, Leuven, Vlaams-Brabant
- France (6):
  - Hopital Lyon Sud, Pierre-Bénite, Auvergne-Rhône
  - Centre Georges Francois Leclerc, Dijon, Bourgogne-Franche-Comté
  - Centre Francois Baclesse (CFB), Caen, Normandy
  - Institut Bergonie, Bordeaux, Nouvelle-Aquitaine
  - Centre Antoine Lacassagne, Nice, Provence Alpes Cote dAzur
  - Institut Gustave Roussy, Villejuif, Île-de-France Region
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Sharet Institute of Oncology, Jerusalem
  - Sheba Medical Center, Tel Litwinsky
- Italy (3):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - Istituto Europeo di Oncologia, Milan
  - Instituto Nazionale Tumori- Fondazione Pascale, Naples
- Netherlands (3):
  - Radboudumc, Nijmegen, Gelderland
  - Erasmus MC, Rotterdam, South Holland
  - University Medical Center Groningen, Groningen
- South Korea (5):
  - Yonsei University Health System, Seoul
  - Asan Medical Center, Univ. of Ulsan, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Spain (8):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Institut Catala dOncologia Badalona, Badalona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Catala d'Oncologia, Barcelona
  - Clinica Universidad Navarra (CUN) Madrid, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario San Carlos, Madrid
  - Hospital Clinico Universitatio Santiago de Compostela, Santiago de Compostela
- United Kingdom (7):
  - University of Oxford, Oxford, Oxfordshire
  - Royal Marsden Hospital - Sutton, Sutton, Surrey
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - University College London Hospitals, London
  - Guys Hospital, London
  - Imperial College Healthcare NHS Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/